CLINICAL TRIAL: NCT00784511
Title: Vitamin D, Glucose Control and Insulin Sensitivity in African-Americans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Susan Harris, Scientist I, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8095; ADA 7-08-CR-27
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; vitamin D; African Americans; overweight; insulin sensitivity; glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Overweight; Insulin Resistance | interventions — Cholecalciferol; Vitamin D; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 vitamin D3 (Experimental): vitamin D3, 4000 IU/d
  Interventions: Dietary Supplement: cholecalciferol
- 2 (Placebo Comparator): placebo
  Interventions: Other: microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: cholecalciferol — 4000 IU/d
  Other Names: vitamin D3; vitamin D
  Arms: 1 vitamin D3
Other: microcrystalline cellulose — 1/d
  Other Names: placebo
  Arms: 2

SUMMARY:
North American blacks tend to have low blood levels of vitamin D because pigmentation blocks vitamin D production in the skin. They also have higher rates of developing type 2 diabetes and higher rates of complications from the disease compared with whites. Although there is compelling evidence that adequate vitamin D may reduce the risk for type 2 diabetes in whites, recent evidence from a national survey demonstrated an association of vitamin D with diabetes in whites but not in blacks. However, the central hypothesis of this study is that providing enough supplemental vitamin D to blacks (raising their blood levels higher than that of most participants in the survey) will improve blood measures related to diabetes risk. The proposed study is a 12-week randomized, double-blind, placebo-controlled experiment designed to examine the effect of vitamin D supplementation (100 μg/d ) on insulin secretion, insulin sensitivity and glucose control in pre-diabetic black men and women aged 40 and older.

ELIGIBILITY:
Inclusion Criteria:

* African-American by self designation
* Glucose intolerance defined as FPG ≥ 100 mg/dl or A1c ≥ 5.8%
* BMI 25.0-39.9
* Age 40 or older

Exclusion Criteria:

Medical Conditions

* Diabetes potentially requiring pharmacotherapy, defined as A1c > 7%
* Uncontrolled thyroid disease
* Current parathyroid, liver or kidney disease
* Renal stone within 5 years
* Sarcoidosis, current pancreatitis, active tuberculosis, hemiplegia, gout
* Inflammatory bowel disease, colostomy, malabsorption
* Cancer other than basal cell skin cancer within 5 years
* Uncontrolled arrhythmia in past year
* Albinism or other condition associated with reduced skin pigmentation
* Pregnancy over the last 1 year
* Intent to become pregnant
* Menopause onset within 1 year
* Any other unstable medical condition Laboratory Tests
* Fasting plasma glucose < 100
* Hemoglobin A1c > 7%
* Laboratory evidence of liver disease (e.g. AST > 70 U/L or ALT > 72 IU/L)
* Laboratory evidence of kidney disease (e.g. estimated glomerular filtration rate < 60 ml/min/1.73 m2).
* Elevated spot urine calcium to creatinine ratio > 0.38 mg/dl*
* Abnormal serum calcium (serum calcium > 10.5 mg/dl)
* Anemia (Hematocrit < 36% in men, <33% in women) Medications (use in past three months)
* Estrogen or testosterone
* Prescription vitamin D
* Lithium
* Oral corticosteroids
* Anti-seizure medications
* Unstable doses of psychotropics or phenothiazines
* Cholestyramine Supplements (current use - may discontinue after screening)
* Vitamin D supplements, cod liver oil, calcium supplements Other
* Body mass index less <25 or > 39.9
* Consumption of more than 14 alcoholic drinks per week
* Inability to attend all three study visits as scheduled
* Inability to provide written informed consent
* age < 40 years
* not African-American (by self-designation)
* Participation in another research intervention study

  * corresponds to a 24-hour urinary calcium excretion > 400 mg

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Insulin secretion rate | 12 weeks
Insulin sensitivity index | 12 weeks
2-hr post load glucose | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States